CLINICAL TRIAL: NCT03614559
Title: Contemporary Clinical Treatment and Long-term Outcomes in Patient With Coronary Chronic Total Occlusion："Time" is the Success Rate of PCI
Brief Title: Contemporary Clinical Treatment and Long-term Outcomes in Patient With Coronary Chronic Total Occlusion
Acronym: PCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Junbo Ge, chief physician, Shanghai Zhongshan Hospital
Other Study IDs: ZS-FDU-20180501
Record Dates: First submitted 2018-07-29; First posted 2018-08-03 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Percutaneous Coronary Intervention
Keywords: chronic total occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CTO PCI group and non CTO PCI group: CTO PCI group： Succession of CTO revascularization non CTO PCI group： Failure or not tried to revascularization
- Initially attempted and re-attempted: PCI initially attempted group： First time to try to revascularization PCI re-attempted group: Second or more time to try to revascularization
- PCI during China Club or not: PCI during Chronic Total Occlusion Club， China Club : CAG in 2016.11.04 Another group: CAG in other time
- Morning，Afternoon，Night: Morning group:（8:00-12:59） Afternoon group：（13:00-17:59） Night group：（after 18:00）

SUMMARY:
In order to know more about contemporary clinical treatment ,epidemiological characteristics, and long-term outcomes in patients with Coronary Chronic Total Occlusion（CTO）in China, the study through collecting and effective analyzing basic information, cardiovascular characteristics, contemporary clinical treatment , and long-term outcomes of CTO patients ,to describe the relevant risk factors ,the contemporary incidence of CTOs and the success rates of CTO percutaneous coronary intervention (PCI), as well as the complications and long-term outcomes of these patients, to explore the relevant factors which affecting the success rates of PCI therapy and to provide safer and more effective advice for the treatment of CTO.

DETAILED DESCRIPTION:
Study Center : Shanghai Zhongshan Hospital

Study Purpose : Through collecting and effective analyzing basic information, cardiovascular characteristics, contemporary clinical treatment , and long-term outcomes of CTO patients ,to describe the relevant risk factors ,the contemporary incidence of CTOs and the success rates of CTO percutaneous coronary intervention (PCI), as well as the complications and long-term outcomes of these patients, to explore the relevant factors which affecting the success rates of PCI therapy and to provide safer and more effective advice for the treatment of CTO.

Study Design : A Retrospective Observational Study

Study Population Description : All CTO patients who has been diagnosed by coronary angiography in Shanghai Zhongshan Hospital in 2016-08-01 to 2020-12-31

Eligibility Criteria :

Entry Criteria :

1. Age ≥17 years old;
2. Finished coronary angiography(CAG) in Shanghai Zhongshan Hospital;
3. CAG found coronary artery(-ies) was/were total occluded more than 3 months;
4. CAG found the diameter of total occluded coronary artery was more than 2.5cm;

Exclude Criteria:

1. Cardiac arrest; Ventricular fibrillation; Cardiogenic shock; Acute thrombosis in the stent; Acute coronary syndrome;
2. The bridge vessel(-s) was/were not total occluded and coronary artery(-ies) was/were total occluded but not trying to revascularize in CAG of the patient who has gone through coronary artery bypass graft before;
3. The diameter was too small or position was too distal of the total occluded coronary artery;
4. Combined severe hepatic or renal insufficiency;
5. The patient who has history of major surgical, cerebral hemorrhage, severe gastrointestinal bleeding, severe anemia, severe allergies, and other anti-platelet drug contraindications in recent 3 months;
6. Pregnant, lactating women;
7. Suffer from malignant tumor or life expectancy less than 2 years

Sample size :

Collecting all cases of CTO patient who has been diagnosed in 2016-08-01 to 2020-12-31 and comply with entry and exclude standards, the expectation of quantity is about 3000-4000.

Follow up time： 2 years

Information collection:

1. Basic information: name, gender, age, hospital number, contact information;
2. Relevant risk factors: medication history, smoking history, drinking history, history of hypertension, history of diabetes, history of dyslipidemia, history of arrhythmia, history of cerebrovascular disease, history of renal insufficiency, previous coronary CTA, and previous myocardial infarction, previous PCI and time, previous CABG surgery and time;
3. Cardiovascular information: Preoperative and postoperative BNP, preoperative and postoperative cTnT, cardiac ultrasonography and LVEF, total occluded coronary artery, collateral circulation establishment, J-CTO score, Progress score, PCI operation mode, contrast agent usage, and final treatment plan;
4. Follow-up content: short-term results (perioperative-related complications) and 2-year long-term results (cardiac and LVEF, cardiac death, re-hospitalization of acute myocardial infarction, and subsequent CABG surgery)

ELIGIBILITY:
Entry Criteria :

1. Age ≥18 years old;
2. Finished coronary angiography(CAG) in Shanghai Zhongshan Hospital in 2016-08-01 to 2017-07-31;
3. CAG found coronary artery(-ies) was/were total occluded more than 3 months;
4. CAG found the diameter of total occluded coronary artery was more than 2.5cm;

Exclude Criteria:

1. Cardiac arrest; Ventricular fibrillation; Cardiogenic shock; Acute thrombosis in the stent; Acute coronary syndrome;
2. The bridge vessel(-s) was/were not total occluded and coronary artery(-ies) was/were total occluded but not trying to revascularize in CAG of the patient who has gone through coronary artery bypass graft before;
3. The diameter was too small or position was too distal of the total occluded coronary artery;
4. Combined severe hepatic or renal insufficiency;
5. The patient who has history of major surgical, cerebral hemorrhage, severe gastrointestinal bleeding, severe anemia, severe allergies, and other anti-platelet drug contraindications in recent 3 months;
6. Pregnant, lactating women;
7. Suffer from malignant tumor or life expectancy less than 2 years

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All CTO patients who has been diagnosed by coronary angiography in Shanghai Zhongshan Hospital in 2016-08-01 to 2017-07-31.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-05-06 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiac and cerebrovascular events (MACCE） | 2 years after CAG
  MACCE, including any of the following adverse events before hospital discharge: death from any cause, Q-wave myocardial infarction, recurrent symptoms Heart and Vessels requiring urgent repeat target vessel revascularization with PCI or CABG, tamponade requiring either pericardiocentesis or surgery, and stroke.

SECONDARY OUTCOMES:
Quality of life assessment | 2 years after CAG
  Two years after having CAG ， we may talk to patient face to face or by phone to help them finish the Seattle Angina Questionnaire （SAQ），measure the score of SAQ and assess the quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided